CLINICAL TRIAL: NCT01283854
Title: Preventing Gestational Diabetes Mellitus Using a Home-based Supervised Exercise Program During Pregnancy
Brief Title: The Cycle Study: a Study of the Effectiveness of Cycling Exercise in Breaking the Cycle of Pregnancy Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: King Edward Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kym Guelfi, Assistant Professor Kym Guelfi, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1003302_Newnham
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2014-11

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental): Each participant randomised to the exercise group will receive routine, regular antenatal care. In addition, these women will be required to participate in three 60-minute exercise sessions each week, starting at 14 weeks gestation, for a total of 14 weeks (i.e. to be completed by 28 weeks of gestation). All exercise sessions will be home-based and fully supervised by an experienced exercise physiologist.
  Interventions: Behavioral: Supervised home-based exercise
- Control group (No Intervention): Women allocated to the control group will not participate in the home-based exercise program, and will continue their normal physical activity throughout pregnancy. This group will receive routine, regular antenatal care, together with the additional outcome assessments at baseline (14 weeks gestation) and cessation of the study (28 weeks gestation).

INTERVENTIONS:
Behavioral: Supervised home-based exercise — Each participant randomised to the exercise group will be required to participate in three 60-minute exercise sessions each week, starting at 14 weeks gestation, for a total of 14 weeks (i.e. to be completed by 28 weeks of gestation). All exercise sessions will be home-based and fully supervised by an experienced exercise physiologist. The exercise program will be implemented in accordance with the American College of Sports Medicine and the American College of Obstetrics and Gynecology guidelines. All sessions will be conducted on a stationary cycle ergometer.
  Heart rate will be measured continuously during exercise to ensure that the exercise intensity is maintained as prescribed. In addition, blood pressure and rate of perceived exertion will be monitored at 10-min intervals. Perceived exertion will not be allowed to exceed a rating of 14 (i.e. "somewhat hard").
  Arms: Exercise group

SUMMARY:
Gestational diabetes mellitus (GDM) is one of the most common medical complications of pregnancy and has serious health implications for both the pregnant woman and her child. In particular, offspring of mothers with GDM have an increased prevalence of obesity, diabetes and metabolic syndrome, perpetuating serious health consequences in subsequent generations.

Although regular exercise offers numerous benefits for both the mother and her child, its effectiveness in preventing GDM remains to be established. It has been recently shown that regular supervised home-based exercise may attenuate the decline in glucose tolerance in obese pregnant women. This study aims to conduct a single-centred, multi-sited, single-blinded randomised controlled trial examining the effect of 14 weeks of supervised home-based exercise (commenced at 14 weeks gestation) on the recurrence and severity of GDM, along with other aspects of maternal and fetal wellbeing.

Eligible participants (n = 200) will be randomly allocated to an exercise intervention (n = 100) or a control group (n = 100). The exercise intervention will involve three 60-minute home-based, supervised exercise sessions each week. This type of program overcomes many of the barriers to exercise in this population including transportation, child care issues and embarrassment associated with exercising in a public venue. The investigators have already shown this program to be both feasible and warmly accepted by obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* women at 12-13 weeks gestation, with a history of gestational diabetes in a previous pregnancy.

Exclusion Criteria:

* unable to participate in the supervised 14 week home-based exercise program
* less than 18 years of age
* unable to understand the implications of participation in the trial
* women with a multiple pregnancy
* women with pre-existing diabetes (type 1 or 2) or cardiac disease
* women currently engaged in a structured exercise program

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2011-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Diagnosis of gestational diabetes mellitus | After the 14 week intervention period (28 weeks gestation)

SECONDARY OUTCOMES:
Insulin sensitivity and glucose tolerance | Pre and post-intervention (14 and 28 weeks of gestation)
Maternal aerobic fitness levels | Pre and post-intervention (14 and 28 weeks gestation)
Maternal morphology (girths and skinfold measures) | Pre and post-intervention (14 and 28 weeks gestation)
Maternal mental health | Pre and post-intervention (14 and 28 weeks gestation)
Obstetric outcomes (rates of medical intervention during labour, birth weight, newborn anthropometrics and incidence of newborn hypoglycemia) | At time of delivery (approximately 40 weeks gestation)

CONTACTS AND LOCATIONS:
Overall Officials: John Newnham, Principal Investigator — The University of Western Australia; Paul Fournier, Principal Investigator — The University of Western Australia; Kym Guelfi, Principal Investigator — The University of Western Australia; Robert Grove, Principal Investigator — The University of Western Australia; Karen Wallman, Principal Investigator — The University of Western Australia; Dorota Doherty, Principal Investigator — Women and Infants Research Foundation
Locations (1):
- King Edward Memorial Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Background] Ong MJ, Guelfi KJ, Hunter T, Wallman KE, Fournier PA, Newnham JP. Supervised home-based exercise may attenuate the decline of glucose tolerance in obese pregnant women. Diabetes Metab. 2009 Nov;35(5):418-21. doi: 10.1016/j.diabet.2009.04.008. Epub 2009 Sep 10. PMID 19747869
- [Derived] Guelfi KJ, Ong MJ, Crisp NA, Fournier PA, Wallman KE, Grove JR, Doherty DA, Newnham JP. Regular Exercise to Prevent the Recurrence of Gestational Diabetes Mellitus: A Randomized Controlled Trial. Obstet Gynecol. 2016 Oct;128(4):819-827. doi: 10.1097/AOG.0000000000001632. PMID 27607876